CLINICAL TRIAL: NCT02391454
Title: Self-monitoring and Empowering Physical Activity With a SMARTphone Application During or After Cancer Treatment in a 12 Week Follow-up: a Randomized Feasibility Study (SMART-trial)
Brief Title: Self-monitoring Physical Activity With a SMARTphone Application in Cancer Patients: a Feasibility Study (SMART)
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMART-2014
Record Dates: First submitted 2015-03-03; First posted 2015-03-18 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms
Keywords: Neoplasms; Cell Phones; Motor Activity; Feasibility
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): usual care
  Interventions: Other: Usual care
- Group B (Experimental): usual care + RunKeeper app
  Interventions: Device: RunKeeper App; Other: Usual care

INTERVENTIONS:
Device: RunKeeper App — Group B will use the RunKeeper app for 12 weeks to self-monitor PA. In the scope of this study, patients merely have to self-monitor PA (e.g. swimming, biking, hiking, running) by GPS or stopwatch function with RunKeeper. Furthermore, patients are requested to activate the 'training reminder' option in the RunKeeper app, which is explained in the user's manual.
  Arms: Group B
Other: Usual care

SUMMARY:
Rationale: Cancer treatment is increasingly successful, resulting in a rising number of cancer survivors. A substantial number of survivors may experience long-term and late side effects from their cancer treatment. In addition, evidence is accumulating that an active lifestyle positively influences cancer treatment outcome and changes the recurrence rates of the disease. Therefore, physical activity (PA) programs are urgently needed and should be incorporated in current treatment regimens. It is noted though that cancer patients and survivors experience difficulties in remaining physically active. A 'smartphone application' (app) may be an accessible way to counteract these problems. The app 'RunKeeper', founded by Mr. Jason Jacobs, 2008, FitnessKeeper Inc. (RunKeeper) is a free, widely spread and well-known app for self-monitoring PA. Convenient features of RunKeeper are self-monitoring PA with GPS or stopwatch, recording progress, goal setting, and personal records. In this study the investigators aim to determine if the RunKeeper app use improves PA by self-monitoring and empowering PA during or after cancer treatment in comparison with usual care in a 12-week follow-up.

Objective: The primary objective is to identify an improvement in PA as measured by the PASE questionnaire when using the RunKeeper app in comparison with usual care for 12 weeks during or after cancer treatment. The investigators hypothesize that the RunKeeper app might assist in stimulating and improving PA behavior. Secondary objectives are to explore the usability of the RunKeeper app.

Study design: The present study is a single-centre prospective two-armed randomized controlled feasibility study.

Study population: Adult patients diagnosed with cancer currently being treated or under surveillance at the department of Medical Oncology at the UMCG.

Intervention: Patients who give informed consent will be randomized in one of the two study arms; 'Group A', usual care (N=15) or 'Group B', usual care + the RunKeeper app (N=15). Directly after randomization, Group B will be sent a brief user's manual for RunKeeper and requested to install the RunKeeper app. Group B will use the RunKeeper app for 12 weeks to self-monitor PA.

Main study parameters/endpoints: The primary endpoint is to calculate the effect-size of the RunKeeper app use for 12 weeks on PA as compared to usual care as measured by the Physical Activity Scale for the Elderly (PASE) questionnaire. The investigators hypothesize that the RunKeeper app might assist in stimulating and improving PA behavior.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age diagnosed with cancer (regardless of type/taxonomy) at the medical oncology department, UMCG
* Patients undergoing cancer treatment or surveillance
* WHO-performance score ≤1
* Signed informed consent

Exclusion Criteria:

* Inability to read or understand the Dutch language
* Inability to handle or not in possession of a smartphone
* Active user of the RunKeeper app
* Severe cardiac (recent cardiovascular event) or psychiatric disease
* Severe kidney or liver impairment
* Pancytopenia
* Patients following supervised oncologic rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Calculate the effect-size of the RunKeeper app use for 12 weeks on PA as compared to usual care | 12 weeks
  The primary endpoint is to calculate the effect-size of the RunKeeper app use for 12 weeks on PA as compared to usual care as measured by the PASE.

SECONDARY OUTCOMES:
To explore the usability of the RunKeeper app use for 12 weeks. | 12 weeks
  The secondary endpoint is the usability of the RunKeeper app as measured by the System Usability Scale (SUS).
To explore patients' experiences of the usability of the RunKeeper app use for 12 weeks. | 12 weeks
  The secondary endpoint is to identify patients' experiences of the usability of RunKeeper as measured by a semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: A.M.E. Walenkamp, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Ormel HL, van der Schoot GGF, Westerink NL, Sluiter WJ, Gietema JA, Walenkamp AME. Self-monitoring physical activity with a smartphone application in cancer patients: a randomized feasibility study (SMART-trial). Support Care Cancer. 2018 Nov;26(11):3915-3923. doi: 10.1007/s00520-018-4263-5. Epub 2018 May 21. PMID 29785635